CLINICAL TRIAL: NCT00380770
Title: A Prospective Randomized Trial Comparing the Response of HIV Kaposi's Sarcoma (KS) to HAART Versus the Combination of HAART and Chemotherapy (CXT)
Brief Title: HIV/AIDS Kaposis Sarcoma: Comparison of Response to HAART vs HAART Plus CXT
Acronym: KAART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: AIDS Care Research in Africa (Other); National Research Foundation, Singapore (Other Government); AIDS Malignancy Consortium (Network); Cipla Medpro (Industry); Dermatological Society of South Africa (Unknown)
Responsible Party: Dr Anisa Mosam, Department of Dermatology UKZN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H029/02
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2009-03

CONDITIONS: HIV; AIDS; Kaposi's Sarcoma; Human Herpesvirus 8
Keywords: HIV; AIDS; Kaposi's sarcoma; Human herpesvirus 8
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sarcoma, Kaposi | interventions — Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAART alone (Experimental): Arm 1. HAART These patients will be given one tablet twice daily of Triomune® (Cipla, Mumbai) Stavudine 40mg b.d > 60 kg , 30mg bd <60kg Lamivudine 150mg b.d > 50 kg 2mg/kg < 50 kg Nevirapine 200mg b.d ( 200mg daily for first 2 weeks)
  Interventions: Drug: Generic HAART Triomune : d4T, 3TC, NVP
- Combination HAART and chemotherapy (Active Comparator): Arm 2. CTX PLUS HAART. HAART will be given as above. In addition, CTX will be administered at 2 weekly intervals in the Oncology Dept at KEH VIII Hospital and will consist of:- Intramuscular Bleomycin 10 U/m2 ; Intravenous Vincristine 1.4mg/m2 maximum 2mg and Intravenous Doxorubicin 20mg/m2.
  Interventions: Drug: Generic HAART Triomune : d4T, 3TC, NVP and chemotherapy ABV

INTERVENTIONS:
Drug: Generic HAART Triomune : d4T, 3TC, NVP — Triomune® (Cipla, Mumbai) Stavudine 40mg b.d > 60 kg , 30mg bd <60kg Lamivudine 150mg b.d > 50 kg 2mg/kg < 50 kg Nevirapine 200mg b.d ( 200mg daily for first 2 weeks)
  Arms: HAART alone
Drug: Generic HAART Triomune : d4T, 3TC, NVP and chemotherapy ABV — Triomune® (Cipla, Mumbai) Stavudine 40mg b.d > 60 kg , 30mg bd <60kg Lamivudine 150mg b.d > 50 kg 2mg/kg < 50 kg Nevirapine 200mg b.d ( 200mg daily for first 2 weeks) Intramuscular Bleomycin 10 U/m2 ; Intravenous Vincristine 1.4mg/m2 maximum 2mg and Intravenous Doxorubicin 20mg/m2.
  Arms: Combination HAART and chemotherapy

SUMMARY:
Kaposi's sarcoma (KS)is the commonest malignancy associated with HIV/AIDS. Therapy for this cancer, which causes substantial morbidity, is suboptimal in resource poor settings. The reasons for this are: advanced state of immunosuppression when patients present for clinical care, concomitant opportunistic infections, non- availability of antiretroviral therapy (ART), non-availability and toxicity of chemotherapy (CXT), when available, in patients with full blown AIDS, prohibitive costs of bone marrow support and fiscal constraints in resource poor settings.

A recent Cochrane Review assessed the effectiveness of current therapeutic regimens for HIV KS, with a focus on options available in resource poor settings. The major selection criteria for this review were randomized controlled trials for HIV KS in adults. The main conclusions were that data from randomized controlled trials on effective treatments for HIV KS are sparse, particularly among people who are also taking highly active antiretroviral therapy (HAART). Alitretinoin gel is effective for therapy of cutaneous lesions, pegylated liposomal doxorubicin is effective for advanced KS and radiotherapy is effective for treating cutaneous lesions. Apart from the randomized trial of radiotherapy, no trials applicable to developing settings were identified. Therapy of HIV KS in developing countries thus remains unanswered.

The authors concluded that therapies discussed in the review are unlikely to be available or affordable in developing countries where the bulk of HIV infection and KS occur, apart from radiotherapy at a few tertiary centers. However, recent changes in pricing due to the global alliance and access initiatives mean that HAART is likely to be more available and accessible to developing countries in the near future. South Africa now has committed to this at cabinet level and had a task force to address this issue.

HAART has been proposed as therapy for HIV KS on the basis of restoring immune competence and minimizing the HIV tat drive to KS formation. It also improves immunologic control of HHV 8 possibly through interrupting the HIV-1- HHV-8 interaction.

There has been only one randomised trial conducted in Spain which compared HAART to the combination of HAART and CXT. There is to date no prospective, randomised controlled trial which compares the efficacy of HAART to the standard of care in HIV KS in Africa.

DETAILED DESCRIPTION:
DETAILED METHODOLOGY

PRIMARY OBJECTIVES:

1.To compare the clinical response of HIV KS at month 12 in patients treated with HAART alone with those treated with the combination of HAART and chemotherapy (CXT).

SECONDARY OBJECTIVES

1. To monitor safety, tolerance and adverse events associated with each regimen.
2. To compare the impact of each regimen at baseline and months 12 on:

   1. CD4 count
   2. HIV1 viral load in blood
   3. HIV disease progression
3. To compare the impact of each regimen on the patients Quality of life (QOL).
4. To compare the impact of each regimen on the patients adherence to HAART. 5 To measure and compare HHV8 viral load and HHV8 specific CTL responses at baseline and month 12 to each regimen.(in blood and tissue specimens )

DESIGN Prospective, randomized, open- labeled trial

RANDOMISATION Patients first staged into GOOD risk and POOR risk groups according to ACTG criteria. Thereafter 4 digit computer generated numbers after staging which assign patients to HAART alone or HAART plus CXT to ensure that equal numbers of GOOD and POOR risk patients are assigned to each group.

INCLUSION CRITERIA

* Signed informed consent
* Adults > 18 years
* Documented HIV positive status (Confirmed by two ELISAs and HIV-1 RNA testing)
* Willingness to use a barrier method of birth control throughout the course of the study, because of potential drug interactions that make oral contraceptives less effective (for women of childbearing potential) and sexually active males
* Histologically proven
* At least five measurable, previously unirradiated cutaneous lesions must be present which can be used as indicator lesions.
* ECOG performance status 0-2

EXCLUSION CRITERIA

* Pregnancy or breastfeeding
* Fungating tumors of KS
* Symptomatic pulmonary KS
* Symptomatic GI tract KS
* Clinical evidence of peripheral neuropathy
* Clinical evidence of heart disease
* Total neutrophil count of < 1,000u/L, Hemoglobin < 9.0gm/dl or platelet count of < 75,000u/L; serum creatinine > 1.5mgh/dl, direct serum bilirubin > 85 umol/l, AST or ALT > 2.5 time ULN.
* Prior HAART ( to fairly evaluate antiretroviral response and KS response to HAART, patients should be antiretroviral naïve)
* Prior radiation therapy for KS to sites of indicator lesions.
* Prior cytotoxic chemotherapy for KS.
* Concurrent neoplasia requiring cytotoxic therapy.
* Life expectancy of < 3 months.
* Circumstances, which in the opinion of the investigator make it unlikely the patient, can comply with the safety monitoring required for participation in this trial.

INTERVENTION Arm 1. HAART These patients will be given one tablet twice daily of Triomune® (Cipla, Mumbai) Stavudine 40mg b.d > 60 kg , 30mg bd <60kg Lamivudine 150mg b.d > 50 kg 2mg/kg < 50 kg Nevirapine 200mg b.d ( 200mg daily for first 2 weeks)

Arm 2. CTX PLUS HAART HAART will be given as above. In addition, CTX will be administered at 2 weekly intervals in the Oncology Dept at KEH VIII Hospital and will consist of:- Intramuscular Bleomycin 10 U/m2 ; Intravenous Vincristine 1.4mg/m2 maximum 2mg and Intravenous Doxorubicin 20mg/m2.

This regimen will be given at 2 weekly intervals. This will be supplied by the Department of Oncology, KwaZulu Natal Province.

PRIMARY ENDPOINTS

1. Clinical response of KS

   * Clinical photographs taken of marker lesions (5 according to AMC criteria) will be taken at baseline, month 6 and 12.
   * Lesion measurement of 5 marker lesions (as per AMC RKS 02 )(www.amc.uab.edu) will be done at baseline, month 3, month 6, month 9 and month 12. Responses will be categorized as complete response(only with biopsy confirmation), complete clinical response, partial response, stable disease and disease progression according to ACTG criteria.
   * The patients will be assessed by a specialist dermatologist, trained to use the above instruments, and will be the same individual so as to decrease bias introduced with inter-observer variability. We recognize that there is the potential for bias as the study is not blinded and dermatologist will know patient assignment. For that reason, we are using established objective criteria to evaluate response.
   * Biopsies will be performed at baseline, month 6 and month 12 to assist in confirming response and to evaluate HIV and HHV8 tissue viral loads
2. Safety and toxicity by DAIDS Toxicity criteria
3. QOL by EORTC QLQ C30
4. Adherence by 7 day adherence questionnaire Adherence will be measured using a standardized validated self administered questionnaire, which enables review of each medication during previous 7 days and a medication specific and overall adherence score.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adults > 18 years
* Documented HIV positive status (Confirmed by two ELISAs and HIV-1 RNA testing)
* Willingness to use a barrier method of birth control throughout the course of the study, because of potential drug interactions that make oral contraceptives less effective (for women of childbearing potential) and sexually active males
* Histologically proven
* At least five measurable, previously unirradiated cutaneous lesions must be present which can be used as indicator lesions.
* ECOG performance status 0-2

Exclusion Criteria:

* • Pregnancy or breastfeeding

  * Fungating tumors of KS
  * Symptomatic pulmonary KS
  * Symptomatic GI tract KS
  * Clinical evidence of peripheral neuropathy
  * Clinical evidence of heart disease
  * Total neutrophil count of < 1,000u/L, Hemoglobin < 9.0gm/dl or platelet count of < 75,000u/L; serum creatinine > 1.5mgh/dl, direct serum bilirubin > 85 umol/l, AST or ALT > 2.5 time ULN.
  * Prior HAART ( to fairly evaluate antiretroviral response and KS response to HAART, patients should be antiretroviral naïve)
  * Prior radiation therapy for KS to sites of indicator lesions.
  * Prior cytotoxic chemotherapy for KS.
  * Concurrent neoplasia requiring cytotoxic therapy.
  * Life expectancy of < 3 months.
  * Circumstances, which in the opinion of the investigator make it unlikely the patient, can comply with the safety monitoring required for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2003-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical response of KS | 3 monthly
  Responses will be categorized as complete response(only with biopsy confirmation), complete clinical response, partial response, stable disease and disease progression according to ACTG criteria.
Skin: tumour measurements of 5 indicator skin lesions. Assessment of KS as per AMC RKS 02 (www.amc.uab.edu) | 3 monthly
  Measurement of the same 5 marker lesions (as per AMC RKS 02 )will be done at baseline, month 3, month 6, month 9 and month 12. Assessed by bi-directional diameter.
photography of indicator lesions with metric tape in frame | 6 monthly
  Clinical photographs taken of marker lesions (5 according to AMC criteria) will be taken at baseline, month 6 and 12.
Visceral: chest radiograph and endoscopy, where necessary, bronchoscopy | 6 monthly
  done in patients who presented with visceral KS at baseline to monitor the disease

SECONDARY OUTCOMES:
Safety and toxicity by DAIDS Toxicity criteria | as they occur
  DAAIDS toxicity criteria used to assess and measure severity of adverse events
Immunological and virological response to HAART as measured by CD4 and HIV-viral load | 3 monthly
  patients CD4 and VL will be measured 3 monthly to assess immunological and virological control
QOL by EORTC QLQ C30 | 3 monthly
  EORTC QLQ C30 will be used as the tool to assess QOL in subjects
Adherence | monthly
  Adherence by 7 day adherence questionnaire Adherence will be measured using a standardized validated self administered questionnaire, which enables review of each medication during previous 7 days and a medication specific and overall adherence score.

CONTACTS AND LOCATIONS:
Overall Officials: Anisa Mosam, FC Derm,PhD, Principal Investigator — Nelson R Mandela School of Medicine, University of Kwazulu Natal
Locations (1):
- Department of Dermatology, King Edward VIII Hospital, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] Sebitloane HM, Mosam A, Moodley J. Disseminated AIDS-associated Kaposi's sarcoma in pregnancy. S Afr Med J. 2006 Jul;96(7):602-3. No abstract available. PMID 16909181
- [Result] Mosam A, Cassol E, Page T, Bodasing U, Cassol S, Dawood H, Friedland GH, Scadden DT, Aboobaker J, Jordaan JP, Lalloo UG, Esterhuizen TM, Coovadia HM. Generic antiretroviral efficacy in AIDS-associated Kaposi's sarcoma in sub-Saharan Africa. AIDS. 2005 Mar 4;19(4):441-3. doi: 10.1097/01.aids.0000161775.36652.85. PMID 15750399
- [Result] Mosam A, Goga Y, Thejpal R, Cassol E, Page T, Cassol S, Aboobaker J, Coovadia HM. Lymphadenopathy, pneumonia, and HIV--a common trio, an uncommon outcome. Lancet. 2005 Jan 15-21;365(9455):266. doi: 10.1016/S0140-6736(05)17747-2. No abstract available. PMID 15652610
- [Result] Cassol E, Page T, Mosam A, Friedland G, Jack C, Lalloo U, Kopetka J, Patterson B, Esterhuizen T, Coovadia HM. Therapeutic response of HIV-1 subtype C in African patients coinfected with either Mycobacterium tuberculosis or human herpesvirus-8. J Infect Dis. 2005 Feb 1;191(3):324-32. doi: 10.1086/427337. Epub 2004 Dec 22. PMID 15633090
- [Result] Peer FI, Pui MH, Mosam A, Rae WI. 99mTc-MIBI imaging of cutaneous AIDS-associated Kaposi's sarcoma. Int J Dermatol. 2007 Feb;46(2):166-71. doi: 10.1111/j.1365-4632.2006.03001.x. PMID 17269969
- [Derived] Shaik F, Uldrick TS, Esterhuizen T, Mosam A. Health-Related Quality of Life in Patients Treated With Antiretroviral Therapy Only Versus Chemotherapy and Antiretroviral Therapy for HIV-Associated Kaposi Sarcoma: A Randomized Control Trial. J Glob Oncol. 2018 Oct;4:1-9. doi: 10.1200/JGO.18.00105. PMID 30354935